CLINICAL TRIAL: NCT05453617
Title: Effects of Intermitting Eating on Weight-Loss Maintenance and Cardiometabolic Risk Factors in Obese Adults: A Randomized Clinical Trial
Brief Title: Intermittent Eating on Sustaining Weight-loss in Obesity
Acronym: INTEREST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huijie Zhang, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2022-155
Record Dates: First submitted 2022-06-18; First posted 2022-07-12 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Obesity
Keywords: Obesity; Time restricted eating; The 5:2 diet; Weight loss maintenance
MeSH Terms: conditions — Obesity; Intermittent Fasting | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The TRE group (Experimental): Participants in the TRE group will be instructed to eat during a window of 8 h/d (8 am to 4 pm).
  Interventions: Behavioral: Time-restricted eating
- The 5:2 diet group (Experimental): Participants in the 5:2 diet group will be instructed to consume 500-600 kcal/d on fast days and eat ad libitum on feast days.
  Interventions: Behavioral: The 5:2 diet
- Control (No Intervention): Participants in the control group will receive a general lifestyle counseling.

INTERVENTIONS:
Behavioral: Time-restricted eating — Participants in the TRE group will be instructed to eat during a window of 8 h/d (8 am to 4 pm)
  Arms: The TRE group
Behavioral: The 5:2 diet — Participants will be instructed to consume 500-600 kcal/d on fast days and eat ad libitum on feast days.
  Arms: The 5:2 diet group

SUMMARY:
Weight regain after weight loss is a major problem in the treatment of obesity. Two novel types of intermittent fasting recently have received more attention: the 5:2 diet and time-restricted eating (TRE). TRE requires individuals to eat in a specified number of hours per day (typically 4 to 10 hours) without energy intake restriction. The 5:2 diet involves 5 feast days and 2 fast days per week; participants eat ad libitum without restriction on feast days while 25% of energy needs (approximately 500-800 kcal per day) are consumed on fast day. This randomized controlled trial aimed to evaluate the effect of TRE and the 5:2 diet on weight loss maintenance and cardiometabolic risk factors after a low-calorie diet in obese adults over 12 months compared to usual health care.

DETAILED DESCRIPTION:
Weight regain after weight loss is a major problem in the treatment of persons with obesity. Two novel types of intermittent fasting recently have received more attention: the 5:2 diet and time-restricted eating (TRE). TRE requires individuals to eat in a specified number of hours per day (typically 4 to 10 hours) without energy intake restriction. The 5:2 diet involves 5 feast days and 2 fast days per week; participants eat ad libitum without restriction on feast days while 25% of energy needs (approximately 500-800 kcal per day) are consumed on fast day. Preliminary evidence suggests that both TRE and the 5:2 diet have beneficial effects on weight loss and cardioprotection in humans. Whether TRE or the 5:2 diet is an effective approach for weight-loss maintenance remains unknown. This randomized controlled trial aimed to evaluate the effect of TRE and the 5:2 diet on weight loss maintenance and cardiometabolic risk factors after a low-calorie diet in obese adults over 12 months compared to usual health care. All participants who have achieved greater than 5% of weight loss after a 8-week low-calorie-diet induced weight loss phase, will be assigned to one of the three study groups (TRE, the 5:2 diet and control groups) in a 1:1:1 ratio. Participants in the TRE group will be instructed to eat during a window of 8 h/d (8 am to 4 pm) over 12 months. Participants in the 5:2 diet group will be instructed to consume 500-600 kcal/d on fast days and eat ad libitum on feast days. Participants in the control group were instructed to receive usual health care.

ELIGIBILITY:
Inclusion Criteria:

* 1.Man or women aged 18-75 years;
* 2.Body mass index (BMI)of 28.0 to 45.0 kg/m2;

Exclusion Criteria:

* 1. History of HIV, hepatitis B or C (self-report) or active pulmonary tuberculosis;
* 2. Diagnosis of type 1 and type 2 diabetes;
* 3. History of malignant tumors;
* 4. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
* 5. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
* 6. History of severe gastrointestinal diseases or gastrointestinal surgery in the past 12 months;
* 7. History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
* 8. Being a smoker or having been a smoker in the 3 months prior to their screening visit;
* 9. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
* 10. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) ;
* 11. Women who are pregnant or plan to become pregnant;
* 12. Patients who cannot be followed for 24 months (due to a health situation or migration);
* 13. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in body weight over 12 months | Baseline to months 12

SECONDARY OUTCOMES:
Change in body fat composition meassured by DEXA | Baseline to months 12
  Body composition is meassured by dual-energy X-ray absorptiometry scans
Change in waist circumference | Baseline to months 12
Change in body mass index | Baseline to months 12
Change in liver fat | Baseline to months 12
  Liver fat is assessed by liver Fibroscan.
Change in systolic blood pressure | Baseline to months 12
Change in diastolic blood pressure | Baseline to months 12
Change in serum triglycerides | Baseline to months 12
Change in serum total cholesterol | Baseline to months 12
Change in serum LDL-c | Baseline to months 12
Change in HbA1c | Baseline to months 12
Change in insulin sensitivity | Baseline to months 12
  Insulin sensitivity is assessed by HOMA-IR
Change in β cell function | Baseline to months 12
  β cell function is assessed by HOMA-B
Change in arterial stiffness measured by pulse wave velocity | Baseline to months 12
  arterial stiffness is measured by pulse wave velocity (PWV)
Change in depression score measured by the Patient Health Questionnaire-9 | Baseline to months 12
  Depression is measured by the Patient Health Questionnaire-9 (PHQ-9)
Change in quality of sleep score measured by the Pittsburgh sleep quality index | Baseline to months 12
  Quality of sleep is measured by the Pittsburgh sleep quality index (PSQI)
Change in quality of life score measured by the 12-item Short-Form Health Survey Questionnaire | Baseline to months 12
  Quality of life is measured by the 12-item Short-Form Health Survey Questionnaire (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD. PhD., Principal Investigator — Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No